CLINICAL TRIAL: NCT00221078
Title: Restoration of Reaching and Grasping Functions in Stroke Patients Using Functional Electrical Stimulation.
Brief Title: Benefits of Applying Neuroprosthesis for Improving Reaching and Grasping Functions in Stroke Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: M. Popovic, Toronto Rehab Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 88098-0461-RR001; 88098-0461-RR001
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Stroke
Keywords: Cerebrovascular Accident; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Neuroprosthesis — The Compex Motion neuroprosthesis, developed by Drs.R. Popovic and Thierry Keller, and company Compex SA, is a flexible device designed to improve grasping function in both SCI and stroke patients. This multi-channel surface stimulation system for grasping provides both palmar and lateral grasp, and holds a number of advantages over the other existing neuroprostesis.
  Other Names: Functional Electrical Stimulation (FES)

SUMMARY:
Functional electrical stimulation (FES) is a process that uses low intensity electrical pulses generated by an electric stimulator to create muscle contractions. By contracting muscles in a specific sequence, one can generate various body functions such as grasping, walking, and standing. Final goal of the study is to evaluate if FES training when applied early during rehabilitation will help stroke patients to use their hands more effectively after discharge from a rehabilitation facility, compared to those patients who have not received FES training.

DETAILED DESCRIPTION:
Neuroprosthesis are systems that apply functional electrical stimulation to cause muscle contractions. If the muscle contractions are sequenced properly one can generate various functions such as grasping, standing, and walking. Recent studies of others and our pilot study indicate that a neuroprosthesis can be successfully applied as a training device to help stroke patients who have hemiplegic arm to relearn how to reach and grasp various objects. The objective of this research program is to confirm these preliminary results with the broader population of stroke patients, and if successful to propose a method to introduce this rehabilitation treatment into Toronto Rehabilitation Institute, Stroke Unit as a primary intervention for hand function recovery. Specifically, our aim is to1)develop an exercise protocol that uses a neuroprosthesis for reaching and grasping developed by our team in combination with the standard physiotherapy treatments to enhance recovery of hemiplegic arm and hand; and 2) assess qualitatively and quantitatively improvements in the reaching and grasping functions achieved with standard rehabilitation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be motivated to participate in the FES study, and must sign the letter of consent.
* Patients must have hemiplegia and the stroke must be confirmed with a CT scan.
* Patients must understand that the role of this study is to enhance recovery and not to guarantee it.

Exclusion Criteria:

* Patients who is motivated and does not sign the letter of consent.
* Patient who has serious cognitive or psychological impairments.
* Patients who has skin rush, allergy or wounds.
* Alcohol or drug abuse.
* Edema in his/her upper extremity.
* Patients with Shoulder Hand Syndrome
* Global aphasia
* Patients who shows early recovery of the function.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-04; Primary Completion 2005-06 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
REL Hand Function Test | 45 min
Fugl-Meyer Assessment | 30 min

SECONDARY OUTCOMES:
Barthel Index | 25 min
Functional Independence Measure | 25 min
Chedoke-McMaster Stages of Motor Recovery | 30 min

CONTACTS AND LOCATIONS:
Overall Officials: Milos Popovic, Ph.D, Principal Investigator — University of Toronto
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

REFERENCES:
- [Result] Popovic MR, Thrasher TA, Adams ME, Takes V, Zivanovic V, Tonack MI. Functional electrical therapy: retraining grasping in spinal cord injury. Spinal Cord. 2006 Mar;44(3):143-51. doi: 10.1038/sj.sc.3101822. PMID 16130018
- [Derived] Marquez-Chin C, Bagher S, Zivanovic V, Popovic MR. Functional electrical stimulation therapy for severe hemiplegia: Randomized control trial revisited. Can J Occup Ther. 2017 Apr;84(2):87-97. doi: 10.1177/0008417416668370. Epub 2017 Jan 17. PMID 28093928
- See also: Rehabilitation Engineering Laboratory — http://www.toronto-fes.ca